CLINICAL TRIAL: NCT06994312
Title: The Impact of Nafamostat Mesylate on the Prognosis of Patients With Sepsis-Induced Coagulopathy Undergoing Hemofiltration：A Single-Center, Prospective, Randomized Controlled Trial
Brief Title: The Impact of Nafamostat Mesylate on the Prognosis of Patients With Sepsis-Induced Coagulopathy Undergoing Hemofiltration
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Yuting Li 20250430
Record Dates: First submitted 2025-04-30; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-04

CONDITIONS: Sepsis-induced Coagulopathy (SIC)
Keywords: Single-Center, Prospective, Randomized Controlled Trial; sepsis-induced coagulopathy (SIC); Nafamostat Mesylate; Prognosis; Hemofiltration
MeSH Terms: interventions — nafamostat; Sodium Citrate; Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nafamostat Mesylate Group (Experimental): Nafamostat mesylate (50 mg/vial, Jiangsu DuRui Pharmaceutical Co., Ltd.) is dissolved and prepared with 5% glucose injection solution. It is continuously infused through the anticoagulant injection tube at the start of hemofiltration, with an initial dose generally ranging from 20 to 50 mg/h. Monitoring is performed before treatment and within 2 to 4 hours after the start of treatment. In cases of active bleeding, moderate to high bleeding risk, hypercoagulable state, or high-dose use of nafamostat mesylate (NM), the monitoring frequency should be increased (e.g., every 4 to 6 hours). After the treatment becomes stable, the monitoring interval can be extended to 12 to 24 hours. The activated clotting time (ACT) or activated partial thromboplastin time (APTT) at the post-dialyzer or venous end should be maintained at 1.5 to 2.5 times the pre-treatment level, or the ACT should be maintained between 150 and 250 seconds, and the APTT between 50 and 70 seconds.
  Interventions: Drug: Nafamostat Mesylate
- Sodium Citrate Group (Active Comparator): Patients were continuously infused with sodium citrate (200 ml/bag, Chengdu Qingshanlikang Pharmaceutical Co., Ltd.). The initial pump rate of 4% sodium citrate was set at 2.1% of the blood flow rate, and the initial pump rate of 10% calcium gluconate was set at 7.3% of the flow rate of 4% sodium citrate. Adjust the doses of sodium citrate and calcium gluconate based on the levels of ionized calcium in arterial and venous blood gases.The goal is to maintain arterial blood ionized calcium levels at 1.00-1.20 mmol/L and venous blood ionized calcium levels at 0.21-0.40 mmol/L.
  Interventions: Drug: sodium citrate

INTERVENTIONS:
Drug: Nafamostat Mesylate — Anticoagulation with Nafamostat Mesylate for SIC Patients Undergoing Hemofiltration
  Other Names: Experimental Group
  Arms: Nafamostat Mesylate Group
Drug: sodium citrate — Anticoagulation with Sodium Citrate for SIC Patients Undergoing Hemofiltration
  Other Names: Control Group
  Arms: Sodium Citrate Group

SUMMARY:
In sepsis, the body is prone to coagulation system disorders, which may progress to sepsis-induced coagulopathy (SIC). When SIC is persistent and cannot be corrected, it often sequentially develops into disseminated intravascular coagulation (DIC) with multiple organ failure. Nafamostat mesylate can be used as an anticoagulant during blood purification in critically ill patients and is also used to treat SIC.Safe and effective anticoagulation is a prerequisite for the success of blood purification therapy. For patients with active bleeding or at risk of bleeding, how to achieve extracorporeal anticoagulation without affecting the body's coagulation function is a major clinical challenge. Nafamostat mesylate can reduce the risk of bleeding during blood purification, but its impact on the survival outcomes of patients with SIC undergoing blood purification therapy remains unclear.The aim of this study is to evaluate the impact of nafamostat mesylate treatment on the prognosis of patients with sepsis-induced coagulopathy undergoing hemofiltration.

ELIGIBILITY:
Inclusion Criteria:

* Adults (Age ≥ 18 years);
* Patients with SIC Undergoing Hemofiltration.

Exclusion Criteria:

* Individuals under the age of 18, pregnant women, and breastfeeding mothers;
* Patients with a history of high sensitivity to nafamostat mesylate (those who have experienced significant bleeding complications from previous use of nafamostat mesylate);
* Fibrinogen < 1.5 g/L;
* Patients with bleeding or high risk of bleeding:

Those in the acute phase of trauma or with active bleeding (e.g., flail chest, obvious contusions of the lungs, liver, spleen, retroperitoneal bleeding, pelvic fractures, etc.); Those with a history of severe head trauma, intracranial surgery, stroke, cerebral aneurysm, or arteriovenous malformation within one month prior to enrollment; Those with a history of congenital bleeding disorders: such as hemophilia; Those with underlying fulminant hepatitis, decompensated cirrhosis, or other severe liver diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
ICU Mortality Rates | Through study completion, an average of 1 year
  The proportion of patients who died during the ICU stay out of the total number of patients in the group.

SECONDARY OUTCOMES:
Average Filter Lifespan | Through study completion, an average of 1 year
  The total sum of all filter usage times for each patient divided by the number of filters used.
ICU length of stay | Through study completion, an average of 1 year
  Length of Stay in the ICU
28-day mortality | Through study completion, an average of 1 year
  The proportion of patients who died within 28 days out of the total number of patients in the group.
Incidence of Bleeding | Through study completion, an average of 1 year
  The proportion of patients experiencing bleeding events (such as cerebral hemorrhage, gastrointestinal bleeding, etc.) during the ICU stay out of the total number of patients.

IPD SHARING:
Plan to Share IPD: No